CLINICAL TRIAL: NCT04705285
Title: Erbium:Yag Laser Versus Pelvic Floor Training for the Treatment of Women With Mild to Moderate Stress Urinary Incontinence: a Pilot Randomized Controlled Trial
Brief Title: Erb:Yag Laser Versus Pelvic Floor Training for the Treatment of Women With Mild to Moderate Stress Urinary Incontinence
Acronym: EFFECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11145
Record Dates: First submitted 2020-08-01; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erbium:Yag Laser (Experimental): Patients allocated to the erbium:yag laser are going to undergo 2 sessions of vaginal laser, separated by one month each other.
  Interventions: Device: Erbium Yag Laser
- Pelvic floor training (Active Comparator): Patients allocated to pelvic floor training, are goin to undergo 10 sessions of pelvic floor exercises coached by an expert physiotherapist.
  Interventions: Behavioral: Pelvic Floor Training

INTERVENTIONS:
Device: Erbium Yag Laser — Subjets in the laser arm will undergo 2 sessions of vaginal erbium-yag laser, separated by a month
  Arms: Erbium:Yag Laser
Behavioral: Pelvic Floor Training — Patients allocated to pelvic floor training, are goin to undergo 10 sessions of pelvic floor exercises coached by an expert physiotherapist
  Arms: Pelvic floor training

SUMMARY:
This is a pilot study to assess the feasibility and safety to run a randomized controlled trial that compared the effectivity of erbium:yag vaginal laser versus pelvic floor training in women with mild to moderate stress urinary incontinence.

DETAILED DESCRIPTION:
This pilot study attempts to demonstrated the feasibility and security to run a randomized controlled study that compared the effectivity of erbium:yag laser used vaginally versus pelvic floor training, coached by a physiotherapist expert in pelvic floor disorders.

Patients are going to be randomized to pelvic floor exercises (10 sessions) or erbium:yag laser (2 sessions), and assess the results at 6 and 12 moths later on.

ELIGIBILITY:
Inclusion Criteria:

* Mild to Moderated Stress Urinary Incontinence

Exclusion Criteria:

* Mixed Urinary incontinence
* Pelvic organ prolase greater than stage 2
* Previous surgery for stress urinary incontinence and/or pelvic organ prolapse
* Severe Stress urinary incontinence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-06-21 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life | The questionnaire will be applied at baseline, 6 month and 1 year
  In order to measure quality of life, we are going to use the International Consultation on Incontinence Questionnaire Short Form (ICQI-SF), validate to spanish and in Chile. A higher score in this scale means a worse outcome for the patient.

SECONDARY OUTCOMES:
Pad test | at baseline, 6 month and 1 year
  A 24 h Pad test will be applied. The pad will be weighted after 24 h of use and the difference between the dry pad and the wet pad is going to be recorded. A great difference means a worse outcome for the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico de La Florida, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No